CLINICAL TRIAL: NCT02618460
Title: Non-contrast Enhanced MR Imaging of the Kidney in Healthy Volunteers
Brief Title: Renal NCE-MRI in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: EC-DG Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Renal NCE-MRI in volunteers
Record Dates: First submitted 2015-11-20; First posted 2015-12-01 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Non-contrast enhanced MRI; healthy volunteers; renal diffusion; renal perfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Whole Group (Experimental)
  Interventions: Device: Non contrast-enhanced magnetic resonance imaging

INTERVENTIONS:
Device: Non contrast-enhanced magnetic resonance imaging

SUMMARY:
Non-contrast enhanced (NCE) structural MRI enables to investigate renal anatomy.

Additional NCE-MR acquisition modalities (e.g. Diffusion Weighted Imaging (DWI), Blood Oxygenation Level Dependent (BOLD) MRI, Arterial Spin Labeling (ASL), MR Angiography (MRA), phase-contrast MRI), which could be used in combination with structural MRI in a single acquisition session, have been identified to investigate in more detail renal function and structure, opening the possibility to estimate local renal diffusion and blood perfusion, beyond providing high-resolution anatomical accuracy.

Preliminary to the identification of novel imaging biomarkers of renal disease progression, perfusion and diffusion MR sequences need to be optimized for the renal compartment. Moreover, NCE-MRIs acquired on healthy volunteers are required to investigate perfusion and diffusion changes in pathological kidneys as compared to normal and physiological condition.

The objective of this study is to provide normal control NCE-MRI sequences to be used as reference for the investigation of perfusion and diffusion changes in the kidney of patients affected by chronic kidney disease (e.g. diabetic nephropathy, nephrosclerosis, autosomal dominant polycystic kidney disease).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 and ≤59 years ;
* Healthy volunteers;
* Written informed consent.

Exclusion Criteria:

* Ferro-magnetic prosthesis, aneurysm clips, severe claustrophobia or other contraindications or exclusions interfering with the MRI assessment;
* Pregnancy (due to safety reasons).

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Apparent Diffusion Coefficient (ADC) | At baseline.
  Renal perfusion and diffusion parameter assessed by Diffusion Weighted Imaging (DWI) MRI, characterising normal physiology.
T2* | At baseline.
  Renal blood oxygenation parameter assessed by Blood Oxygenation Level Dependent (BOLD) MRI, characterising normal physiology.
Renal artery flow. | At baseline.
  Renal perfusion parameter assessed by Phase-Contrast (PC) MRI, characterising normal physiology.

CONTACTS AND LOCATIONS:
Locations (1):
- Unità di Nefrologia e Dialisi - A.O. Papa Giovanni XXIII, Bergamo, Bergamo, Italy